CLINICAL TRIAL: NCT06383819
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Parallel-group Study to Evaluate the Efficacy and Safety of Longidaza® for the Treatment of Patients With Residual Changes in the Lungs After COVID-19
Brief Title: Efficacy and Safety of Longidaza® for the Treatment of Patients With Residual Changes in the Lungs After COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Long-Cov-III-21
Record Dates: First submitted 2024-04-24; First posted 2024-04-25 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Post-Acute COVID-19 Syndrome; Lung Disease With Polymyositis; Fibrosis; Lung Diseases, Interstitial; Lung; Disease, Interstitial, With Fibrosis
Keywords: Lung Diseases; COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fibrosis; Lung Diseases, Interstitial; Disease; Lung Diseases; COVID-19 | interventions — Longidaza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Longidaza® (Experimental): Bovhyaluronidase azoximer, 3000 IU
  Interventions: Drug: Longidaza®
- Placebo (Placebo Comparator): The placebo will contain no active pharmaceutical ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Longidaza® — dose 3000 IU intramuscularly once every 5 days, 15 injections
  Other Names: Bovhyaluronidase azoximer
  Arms: Longidaza®
Drug: Placebo — intramuscularly once every 5 days, 15 injections
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to evaluate the efficacy and safety of Longidaza®, lyophilisate for preparation of solution for injection, at a dose of 3000 IU compared to placebo in the treatment of adult patients with residual changes in the lungs after COVID-19 infection

DETAILED DESCRIPTION:
The main objective of the clinical study was to prove the superiority of the efficacy of the drug Longidaza® over placebo when used in adult patients with residual changes in the lungs after COVID-19 infection based on the dynamics of respiratory function

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 to 80 years, who signed an informed consent form.
2. The condition after infection with COVID-19, documented in the period from 1 to 12 months before screening (ICD-10: U07.1, U07.2), including accompanied by hospitalization of the patient.
3. The presence of a negative result of the polymerase chain reaction test (PCR) during screening and an express test for the SARS-CoV-2 antigen at visit 2.
4. The presence of respiratory symptoms (at least dyspnea), while the severity of dyspnea on the mMRC during screening is ≥ 1 point.
5. The value of hemoglobin oxygen saturation: SpO2 < 95% at rest at the screening; and/or desaturation (decrease of SpO2 by ≥ 4% in the 6MWT relative to the value at rest) at the screening.
6. The presence of residual changes in the lung parenchyma characteristic of previous COVID-19 infection, > 10% of the area, according to CT at the screening
7. Respiratory dysfunction of the restrictive type at the screening: FVC < 80%, FVC 1 / FVC > 70%.

Exclusion Criteria:

1. A history of chronic respiratory diseases (interstitial lung disease, chronic obstructive pulmonary disease, bronchial asthma, bronchiectasis, lung cancer).
2. Clinical signs or anamnesis data on the presence of diseases that, according to the researcher, can lead to restrictive changes in respiratory function (pronounced kyphoscoliosis, pleural effusion, neuromuscular diseases), pathological obesity, etc.
3. Clinical signs or anamnesis data on the presence of unstable angina pectoris, stable angina pectoris of high functional class, clinically significant cardiac arrhythmias, chronic heart failure, pulmonary hypertension, suffered pulmonary embolism or acute myocardial infarction in within 6 months prior to screening.
4. Dyspnea of any other etiology: thyrotoxicosis, anemia (hemoglobin less than 100 g/l), pathological obesity (BMI ≥ 40 kg/m2), metabolic acidosis, neuromuscular diseases according to anamnesis or screening examination.
5. The presence of an acute infectious process of any etiology and localization.
6. Allergic reactions to the administration of azoximer bovhyaluronidase or an auxiliary component of the studied drug (mannitol) in the anamnesis.
7. Clinical signs of pulmonary hemorrhage and/or hemoptysis during examination and in the anamnesis.
8. Confirmed eye injuries with vitreous hemorrhage during the last 6 months according to the medical history.
9. Malignant neoplasms of any localization in the anamnesis, with the exception of in situ carcinoma, which required only surgical treatment.
10. Renal failure.
11. Taking drugs of prohibited therapy since the start of screening in this study.
12. Serological test positive for HIV infection, viral hepatitis B and C.
13. Pregnancy or breastfeeding.
14. Participation in clinical trials of an experimental drug within 30 days prior to screening for participation in the current study.
15. Any other medical or social conditions that, in the opinion of the research physician, do not allow the patient to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Forced vital capacity (FVC) (visit 4) | Baseline to Day 71±1
  Change in the FVC (%) compared with the initial data according to spirometry data after completion of the course of therapy

SECONDARY OUTCOMES:
Slowing the decline in respiratory function | Baseline to Day 180±3
  Slowing the decline in respiratory function (FVC (%) compared with the initial data after the end of the observation period
Change in FVC (visit 5) | Baseline to Day 180±3
  Change in the FVC (%) compared with the initial data after the end of the observation period
The proportion of patients with an increase in the FVC (%) | Baseline, Day 71±1, Day 180±3
  The proportion of patients with an increase in the FVC (%) by 10% or more compared to the initial values after Visit 4 and Visit 5
Dynamics of hemoglobin oxygen saturation (SpO2) | Baseline, Day 71±1, Day 180±3
  Dynamics of SpO2 values at rest after Visit 4 and Visit 5
The proportion of patients with SpO2 ≥ 93% and < 93% | Baseline, Day 71±1, Day 180±3
  The proportion of patients with SpO2 value at rest ≥ 93% and < 93% after Visit 4 and Visit 5
The proportion of patients with desaturation | Baseline, Day 71±1, Day 180±3
  The proportion of patients with desaturation, defined as a decrease in SpO2 by ≥ 4% after 6-minute walk test (6MWT) after Visit 4 and Visit 5
The proportion of patients with an increase in the distance of 6MWT | Baseline, Day 71±1, Day 180±3
  The proportion of patients with an increase in the distance of 6MWT by 50 m or more after Visit 4 and Visit 5
The proportion of patients with a decrease in the severity of dyspnea on the Borg scale | Baseline, Day 71±1, Day 180±3
  The proportion of patients with a decrease in the severity of dyspnea on the Borg scale by ≥ 2 points after Visit 4 and Visit 5
The proportion of patients with a decrease in the severity of dyspnea on the Modified Medical Research Council Dyspnea Scale (mMRC) | Baseline, Day 71±1, Day 180±3
  The proportion of patients with a decrease in the severity of dyspnea on the mMRC by ≥ 1 point after Visit 4 and Visit 5
Change in cough severity on the Visual Analogue Scale (VAS) | Baseline, Day 71±1, Day 180±3
  Change in cough severity on the VAS after Visit 4 and Visit 5
Change in the assessment of the quality of life according to the European Quality of Life 5-Dimension 5-Level Questionnaire (EuroQol-5D-5L) | Baseline, Day 71±1, Day 180±3
  Change in the assessment of the quality of life according to the EuroQol-5D-5L after Visit 4 and Visit 5

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Avdeev, DM, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (30):
- Russia (30):
  - State Autonomous Healthcare Institution of the Sverdlovsk region "Aramil City Hospital", Aramil
  - Private healthcare institution "Clinical Hospital "RZD-Medicine" of the city of Chelyabinsk", Chelyabinsk
  - State Budgetary Healthcare Institution "Regional Clinical Hospital No. 3", Chelyabinsk
  - Alliance Biomedical-Ural Group LLC, Izhevsk
  - Federal State Budgetary Educational Institution of Higher Education "Kazan State Medical University" of the Ministry of Health of the Russian Federation. The State Autonomous healthcare institution "Hospital for War Veterans of Kazan", Kazan'
  - Federal State Budgetary Educational Institution of Higher Education "Kazan State Medical University" of the Ministry of Health of the Russian Federation, Kazan'
  - State Autonomous Healthcare Institution "Kuzbass Clinical Hospital of Emergency Medical Care named after M.A. Podgorbunsky", Kemerovo
  - Medical Center Rhevma-Med LLC, Kemerovo
  - Federal State Budgetary Educational Institution of Higher Education "Kirov State Medical University" of the Ministry of Health of the Russian Federation, Kirov
  - Federal State Budgetary Institution "National Medical Research Center for Therapy and Preventive Medicine" of the Ministry of Health of the Russian Federation, Moscow
  - Federal Budgetary Institution of Science "Central Research Institute of Epidemiology" of the Federal Service for Supervision of Consumer Rights Protection and Human Well-being, Moscow
  - Unimed-S Zao, Moscow
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - ErSi Medical LLC, Novosibirsk
  - Professorial Clinic LLC, Perm
  - Energia Zdoroviya LLC, Saint Petersburg
  - Medical Center Reavita Med SPb LLC, Saint Petersburg
  - Reavita Med SPb Medical Center LLC, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Consultative and Diagnostic Center No. 1"., Saint Petersburg
  - Eco-Safety Research Center LLC, Saint Petersburg
  - Federal State Budgetary Institution "Consultative and Diagnostic Center with Polyclinic" of the Office of the President of the Russian Federation, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "Consultative and Diagnostic Center No.85", Saint Petersburg
  - Astarta LLC, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Saratov State Medical University named after V.I. Razumovsky" of the Ministry of Health of the Russian Federation, Saratov
  - Regional State budgetary healthcare institution "Clinical Hospital No. 1", Smolensk
  - Federal State Budgetary Educational Institution of Higher Education "Siberian State Medical University" of the Ministry of Health of the Russian Federation, Tomsk
  - Budgetary healthcare institution of the Voronezh region "Voronezh Regional Clinical Hospital No. 1", Voronezh
  - Medical Center for Diagnosis and Prevention plus LLC, Yaroslavl
  - The State Autonomous Healthcare Institution of the Yaroslavl region "Clinical Hospital No. 9", Yaroslavl
  - Ural research Institute of Phthisiopulmonology, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No